CLINICAL TRIAL: NCT05217485
Title: Continuous Ambulatory Cardiac Monitoring for Recurrent Atrial Fibrillation After Sepsis
Acronym: CAMS-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Isuru Induruwa, Clinical Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAMSAF
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation; Sepsis; Infections; Cardiac Arrhythmia
Keywords: atrial fibrillation; sepsis; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Sepsis; Infections; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Interventional single arm, prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infection and reverted atrial fibrillation (Experimental): Patients who have developed first-diagnosed atrial fibrillaiton in the context of sepsis or infection
  Interventions: Device: Zio 14-day cardiac patch

INTERVENTIONS:
Device: Zio 14-day cardiac patch — A wearble adhesive cardiac patch (14-day) called Zio

SUMMARY:
To detect atrial fibrillation after infection.

DETAILED DESCRIPTION:
This study will prospectively recruit patients who are admitted to CUH general medical wards due to an infection or sepsis and develop new/first diagnosed transient AF. In CUH, our previous projects have shown that around 1500 patients are admitted under general medicine each month at least 1 new diagnosis of AF is made each day (30/month)26.

In particular to the cohort that develop sepsis, they may well be frail and elderly where anticoagulation is often not prescribed as a result 27 unless definitive diagnosis of recurrent AF would be made. The CAMS-AF study will closely tie in with an already existing stroke prevention service at CUH (SOS-AF) who are already screening for patient admitted with AF on general medical wards and will therefore be able to identify those with new AF during an episode of sepsis. Potential participants will be approached by the study investigators prior to discharge and if they are in sinus rhythm written consent will be obtained to place a non-invasive wearable cardiac monitor patch for 14-days, to detect any subclinical arrhythmias, particularly AF.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Admission with any infection or sepsis
* Transient AF
* Under general medicine
* Can be anticoagulated or not
* Sinus rhythm at discharge or point of Zio patch placement

Exclusion Criteria:

* Previous history of AF or paroxysmal AF
* Age less than 18 years
* Pregnancy
* Active and known malignancy
* Recent cardiac or non-cardiac surgery (3 months)
* Recent myocardial infarction (3 months)
* Individuals with skin allergies to plasters and adhesive devices
* Chest wall deformity, skin condition over sticker site
* History of thyroid disease
* Current alcohol intake above recommended limits
* Already has a cardiac monitor or pacemaker inserted
* Known contraindication for anticoagulation therapy
* Patients who lack capacity or have an estimated life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Quantify the incidence of early (within 14-days) AF recurrence in patients who are being discharged, following hospitalisation for an infection or sepsis and develop transient AF at CUH. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared